

# Follow-up of Phase I/II study of CaspaCIDe T cells (BPX-501) from an HLA-partially matched family donor after negative selection of TCR αβ+T cells in pediatric patients affected by hematological disorders

| Protocol Number: | BP-404 |
|---|---|
| Combination Product: | BPX-501 - Donor T cells genetically modified with BPZ-<br>1001 retroviral vector containing the iCasp safety gene<br>Rimiducid (Dimerizer drug) |
| Principal Investigators and Institutions: | Prof. Franco Locatelli IRCCS Ospedale Pediatrico Bambino Gesù Piazzale Sant'Onofrio, 4 00161 Roma, Italy Dr. Mohammed Fuad M. Essa King Abdullah International Medical Research Centre P.O. Box 3660, Riyadh 11481, Mail Code 1515 (KAIMRC) |
| Trial Sponsor: | Bellicum Pharmaceuticals, Inc.<br>2130 W. Holcombe Blvd, Suite 800<br>Houston, TX 77030 |
| ClinicalTrials.Gov / EudraCT Number: | 2016-003226-16 |
| Version Number: | 4.0 |
| Date: | 30 June 2020 |

# Confidentiality Statement

This document contains information confidential to Bellicum Pharmaceuticals, Inc. and it may not be disclosed to anyone other than recipient study staff and members of Institutional Review Boards (IRBs) and Ethical Committees (ECs). This information cannot be used for any purpose other than either evaluation or conduct of the clinical study described here without prior written consent from Bellicum Pharmaceuticals, Inc.

Version 4.0 

# Investigator's Agreement

I have read this protocol and agree to comply with all provisions set forth in this protocol, including all statements regarding confidentiality, and to complete the study within the time designated.

I assume responsibility for the conduct of this study at my study site. I will ensure that I have sufficient resources allocated to this project such that the safety of my patients is protected at all times and that I complete my obligations to the Sponsor according to the agreed timelines. I will delegate responsibilities only to those who are qualified by training and experience. I will ensure the integrity of the data generated by my team and that all team members are familiar with the study protocol and the study medication.

I agree that I will grant access to the applicable records, my staff allocated to the conduct of this protocol and my facilities for the purposes of monitoring, auditing and any required inspections associated with the conduct of this clinical trial.

I agree to comply with the ICH Guideline on Good Clinical Practice, applicable EMA regulations and applicable FDA guidelines set forth in 21 CFR Parts 11, 50, 54, 56, and 312.

Confidential information contained in the protocol document will not be used for any other purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of the Sponsor.

| Signature | Date |
|--------------|------|
| Printed Name | |
| Investigator | |


# SIGNATURES AND AGREEMENT WITH THE PROTOCOL

| - | | | | 4.7 | |
|---|---|-----|-----|-----|----|
| 1 | ľ | toc | nI. | tl | ٥. |

Follow-up of Phase I/II study of CaspaCIDe T cells (BPX-501) from an HLA-partially matched family donor after negative selection of TCR  $\alpha\beta$ +T cells in pediatric patients affected by hematological disorders

# Sponsor Approval

Sponsor: Bellicum Pharmaceuticals Inc.

| I have reviewed | and approved the | protocol and con | firm that the | protocol | follows G( | CP. |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

| Signature: | Date: |
|-----------------------------------------------------|-------|
| Name: Charity Scripture, MS, PharmD, BCOP | |
| Title: Vice President, Clinical and Medical Affairs | |


# TABLE OF CONTENTS

| Investigator's Agreement | 2 |
|------------------------------------------------------------------|----|
| SIGNATURES AND AGREEMENT WITH THE PROTOCOL | 3 |
| TABLE OF CONTENTS. | 4 |
| 1 BACKGROUND | 6 |
| 2 SYNOPSIS | 7 |
| 3 LIST OF ABBREVIATIONS AND TERMS | 10 |
| 4 INTRODUCTION | 12 |
| 4.1 BPX-501: Genetically Modified T Cells With Safety Switch | 12 |
| 4.2 Evaluation of Benefits/Risks | 14 |
| 5 OBJECTIVES OF THE STUDY | 14 |
| 5.1 Primary Objective | 14 |
| 5.2 Secondary Objectives | 14 |
| 5.3 Estimated Enrollment | 14 |
| 5.4 Subject Inclusion Criteria | 14 |
| 5.5 Subject Exclusion Criteria | 15 |
| 6 PATIENT POPULATION AND SELECTION | 15 |
| 6.1 Patient Discontinuation/Withdrawal Criteria | 15 |
| 7 DESIGN AND CONDUCT OF THE STUDY | 16 |
| 7.1 Trial Rationale | 16 |
| 7.2 Trial Design | 17 |
| 7.3 Patient Enrollment, Registration and Assignment to Treatment | 17 |
| 7.4 Rimiducid Dimerizer Drug Packaging, Labeling and Storage | 17 |
| 7.5 Infusion of Rimiducid | 18 |
| 7.6 Monitoring | 19 |
| 7.7 Management of Experimental Drugs | 20 |
| 8 TREATMENTS IN ASSOCIATION WITH SAES EVALUATION | |
| CRITERIA | 20 |

| | 8.1 | Laboratory Investigations | 20 |
|---|---|---|---|
| 9 | RE | ESPONSE AND TOXICITY EVALUATION | 21 |
| | | Parameters of safety, assessment of AE and SAE during the duration of the | 21 |
| | | Expedited Reporting Requirements for Serious Adverse Events | |
| | | End of Study | |
| 10 | | ATA COLLECTION, QUALITY ASSURANCE AND MANAGEMENT | |
| | 10.1 | Recording of Data | 26 |
| | 10.2 | 2 Data Quality Assurance | 26 |
| | 10.3 | B Data Management | 26 |
| | 10.4 | Statistical Methods | 27 |
| | 10.5 | Reporting of Deviations to the Protocol | 29 |
| 11 | ET | THICAL ISSUES/CONSIDERATIONS | 29 |
| | 11.1 | Institutional and Ethical Review | 29 |
| | 11.2 | 2 Investigator's Responsibilities | 30 |
| 12 | RE | FERENCES | 31 |
| A | ppen | dix A: Chronic GVHD Grading Scale and Assessment | 32 |
| A | ppen | dix B: Management of Chronic GVHD (cGVHD) | 39 |
| A | ppen | dix C: Corticosteroid Conversion Table | 41 |
| A | ppen | dix D: AE Grading and Toxicity | 42 |
| A | ppen | dix E: Guidelines for Monitoring & Management of Neurotoxicity | 43 |
| A | ppen | dix F: Assessments Associated with Rimiducid in Treatment of GVHD | 48 |
| Li | st of | f Tables | |
| Ta | ble | 1: Schedule of Events (Laboratory and Clinical) | 8 |
| | | 2: Gene Therapy Monitoring Schedule | |
| Ta | ble | 3: Guidance for Adverse Event Reporting | 22 |


# 1 BACKGROUND

Over the past 4 decades, allogeneic hematopoietic stem cell transplantation (allo-HSCT) from an HLA-matched donor, either related or unrelated, has been increasingly used to treat patients affected by several malignant or non-malignant disorders. However, only 25% of patients who need or could benefit from an allograft have an HLA-identical sibling and fewer than 60% of remaining patients can be matched with suitable HLA-compatible, unrelated donors (Rocha 2008). In the absence of an HLA-matched donor, alternative donor/sources of hematopoietic stem cells such as HLA-haploidentical relatives are being increasingly used. While mature donor T cells present in the graft facilitate T-cell reconstitution, in the context of increased immune genetic disparity between patient and donor, the T cells are also responsible for the occurrence of graft-versus-host disease (GVHD), a severe, sometimes fatal, immune complication, which also impairs patient's immune reconstitution.

Strategies to prevent GVHD after HLA-haploidentical allo-HSCT based on either pharmacological immunosuppression or T-cell depletion of the graft have been developed. In particular, the physical elimination of T cells from the graft has been shown to be highly effective to prevent both acute and chronic GVHD (cGVHD). However, with T- cell depletion of the graft, the patient cannot benefit from the adoptive transfer of donor-derived memory T lymphocytes, which are mainly responsible for protection from severe infections during the state of profound immune deficiency that usually lasts for at least 4-6 months after transplantation. Overall, HLA-haploidentical allo-HSCT is associated with a higher incidence of graft rejection, and both viral and fungal infections, resulting in high transplantation-related mortality (TRM).

US and European gene therapy guidelines require monitoring delayed adverse events in patients who are exposed to gene therapy products for a period of 5-15 years depending on the nature of the product. A potential, but rare, risk of gene therapy using retroviral vectors is the generation of a replication competent retrovirus. This long term follow-up observation period provides a chance to mitigate risks associated with the gene therapy.


# 2 SYNOPSIS

| Study Identifier(s) | DD 404 Feeder CT #2016 002226 16 |
|---|---|
| Study Identifier(s) | BP-404 EudraCT #2016-003226-16 |
| Aim of the Study | This is a Phase I/II study to evaluate the long-term safety of<br>the infusion of BPX-501 gene-modified T cells after<br>mismatched, T cell-depleted allogeneic transplantation and<br>evaluate disease free survival at 1 and 2 years post-transplant |
| G. 1. D. : | Open label, multi-centre, non-randomized, non-controlled long-term safety evaluation |
| Study Design | Follow-up of all patients enrolled on BP-004 and treated with BPX-501 who are beyond Day 180 and have completed or discontinued the parent study. |
| Study Population | The patient population is identical to BP-004 as it is the long-term follow-up of those patients. Estimated enrolment up to 175 BP-004 patients. |
| Main Inclusion Criteria | <ol> <li>Signed written informed consent by the patient or the patient's guardian for children who are minors</li> <li>Enrolled on BP-004 protocol, received BPX-501 infusion, completed or discontinued from the study, and are beyond Day 180.</li> </ol> |
| Main Exclusion Criteria | Lack of parents'/guardian's informed consent for children who are minors Withdrawal from BP-004 study prior to BPX-501 infusion. |
| Dosage, Treatment<br>Regimen, Route of<br>Administration | No BPX-501 infusions will be administered under this protocol. Rimiducid to be given at 0.4 mg/kg weight (intravenous infusion) only in the setting of uncontrolled GVHD. |
| Locations (e.g. regions) | Italy, Saudi Arabia. |
| Primary Endpoint(s) with<br>Time Point(s) of<br>Assessment | Overall Survival and incidence of Disease-Free Survival in<br>both malignant and non-malignant patients at 1 year and 2<br>years post-transplant. Relapse-Free Survival in malignant<br>patients at 1 year and 2 years post-transplant. |
| Main Secondary Endpoint(s) with Time(s) of Assessment | Long-term safety for a total of 15 years from BPX-501 administration |


Table 1: Schedule of Events (Laboratory and Clinical)

| Time - Months (+/-14 Days) | 9 | 12 | 15 | 18 | 21 | 24 | 30 | 36 | 42 | 48 | 54 | 60 | YEARLY | 6-15 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Overall Survival (OS) | | X | | | | X | | X | | X | | X | | X |
| Disease-Free Survival (DFS) | | X | | | | X | | X | | X | | X | | X |
| Relapse-Free Survival (RFS) | | X | | | | X | | X | | X | | X | | X |
| Hematology; Chemistry | X | X | X | X | X | X | | | | | | | | |
| Immune Reconstitution <sup>1</sup> : | X | X | X | X | X | X | | | | | | | | |
| RCR <sup>4</sup> | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Modified History & Physical | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Neurological Exam⁵ | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Vital Signs <sup>2</sup> | X | X | X | X | X | X | | | | | | | | |
| GVHD Assessment <sup>6</sup> | X | X | X | X | X | X | | | | | | | | |
| Concomitant Medication <sup>3</sup> | X | X | X | X | X | X | | | | | | | | |
| Adverse Event | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Bellicum Research Samples | Research samples (peripheral blood and/or tissue) for assessment of BPX-501 cells (CD3+CD19+) will be collected and sent to the sponsor prior to administration of systemic corticosteroids doses (e.g. methylprednisolone), at 4-hours (± 30 minutes) and 24-hours (± 1 hour) | | | | | | | | | | | | | |
| Rimiducid Infusion <sup>7</sup> | post-systemic corticosteroid initiation, and at 7-days, 14-days, 21-days, and 28-days (± 24 hours) post-systemic corticosteroid initiation. BPX-501 Cellular Kinetics (post-rimiducid) Within 4 hours (± 30 minutes) prior to initiation of rimiducid infusion, 30 minutes), then at 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, and 24 hours (± 30 minutes) after initiation of infusion (of each dose of rimiducid) samples will be collected (and will be split for separate processing). Subsequently at 48 hours (± 1 hour) and 7 days (after initiation of infusion of each dose of rimiducid), and then at 14 days, 21 days, and 28 days (± 24 hours) after the final dose of rimiducid (if more than one dose is administered) blood samples will be drawn and evaluated for T cell responses only. Rimiducid Pharmacokinetics (PK): As achievable, blood samples will be drawn at the following time-points (in the same series as the split samples above): within 4 hours (± 30 minutes) prior to the initiation of rimiducid infusion; 30 mins (± 5 minutes) after initiation of the infusion; at 2 hours (< 5 min prior to end of the rimiducid infusion), 4 hours, 6 hours, 8 hours, 12 hours, and 24 hours (± 30 minutes) after the start of the infusion. (see Appendix F). | | | | | | | | | | | | | |


- 1 Peripheral blood (~12 mL, in green top tubes; as feasible for patient weight) shall be collected for Immune Reconstitution and clinical flow cytometry studies. The basic clinical flow panel includes CD3+ cells, (if achievable, alpha/beta CD3+ cells, gamma/delta CD3+ cells), CD4+ cells, CD8+ cells, Natural Killer cells, B cells, and CD3+/CD19+ cells, CD3+/CD19+/CD4+ cells and CD3+/CD19+/CD8+ cells. Additional flow panels may be included as deemed necessary by the treating physician. IgG, IgM and IgA levels shall be reported.
- 2 Vital signs include blood pressure, heart rate, respiratory rate and temperature.
- 3 Concomitant Medication: The protocol will be conducted during the routine clinical care of the patients. All treatments and critical medications, defined below shall be collected in the EDC database:
- Treatment for GVHD
- · Prophylaxis and/or treatment for infectious complications
- · Treatments in association with serious adverse events (SAE)s

Standard supportive care treatments, non-prescription medications/OTCs, NSAIDs, laxatives/stool softeners, vitamins, and herbal supplements will not be collected if they are not protocol-mandated.

- 4 Two purple top tubes (heparinized) of whole blood to be collected and frozen and then batch shipped to the Sponsor or designee per instructions in the laboratory manual for collection of the gene therapy monitoring.
- 5 For clinical assessment and management of neurotoxicity refer to Appendix E.
- 6 GvHD assessments will be performed according to standard practice in the hospital. Refer to Appendix A and Appendix B.
- 7 Research blood sample collection for rimiducid infusion to be sent as directed. Refer to Appendix F for collection and processing of samples for pPK testing.

Version 3.0 

# 3 LIST OF ABBREVIATIONS AND TERMS

AE Adverse Event

aGVHD Acute Graft Versus Host Disease

Allo-HSCT Allogeneic hematopoietic stem cell transplantation

CFR Code of Federeal Regulations

cGVHD Chronic Graft Versus Host Disease

CNS Central Nervous System

CRF Case Report Form

CRO Contract Research Organization

CTL Cytotoxic T Lymphocytes

DFS Disease Free Survival

eCRF Electronic Case Report Form

DEHP Bis(2-ethylhexyl) phthalate

EC Ethics Committee

EDC Electronic Data Capture

EMA European Medicines Agency

FDA Food and Drug Administration

FKBP Human FK-506-binding protein

GCP Good Clinical Practice

GI Gastrointestinal

GVHD Graft Versus Host Disease

HLA Human Leukocyte Antigens

HSV Herpes Simplex Virus

iCasp 9 Inducible Caspase 9

ICH International Conference on Harmonization

IMP Investigational Medicinal Product

IRB Institutional Review Board

IV Intravenous

LTFU Long-term Follow Ups

NCI CTCAE National Cancer Institute Common Terminology for Adverse Events


NGHA Ministry of Naional Guard – Health Affairs

NSAID Nonsteroidal Anti-inflammatory Drugs

OPBG Ospedale Pediatrico Bambino Gesù

OTC Over the Counter

PCR Polymerase Chain Reaction

PD Pharmacodynamics

PK Pharmacokinetics

pPK Population PK

RFS Relapse-Free Survival

RCR Replication Competent Retrovirus

SAE Serious Adverse Event

SUSAR Serious Unexpected Serous Adverse Reaction

TCR T-Cell Receptor

TK Thymidine Kinase

TRM Transplant-Related Mortality

VCN Vector Copy Number


# 4 INTRODUCTION

# 4.1 BPX-501: Genetically Modified T Cells With Safety Switch

# 4.1.1 iCasp9 Safety Gene

Unmodified donor T cell infusion is potentially an effective strategy for conferring anti-viral and anti-tumor immunity following allo-HSCT (Di Stasi 2011). However, the administration of greater than 10<sup>5</sup> cells/kg unmodified donor T cells to recipients of haploidentical stem cell transplantation has been associated with increased incidence of GVHD. It has been previously demonstrated that administration of up to 10<sup>7</sup> cells/kg of CD25+ allodepleted donor T cells after haploidentical transplantation for hematological malignancies could be administered safely and that the addition of these T cells was effective in controlling viral disease (Amrolia 2006). However, mortality due to disease relapse remained high, presumably due to the fact that the estimated frequency of tumor-reactive precursors is 1 to 2 logs lower than the frequency of virus- reactive precursors.

The use of higher numbers of allodepleted T cells containing an inducible caspase 9 safety gene in order to treat the potential increase in GVHD was then evaluated. The caspase recruiting domain of the human caspase 9 was modified with a drug binding domain, permitting T cell elimination after administration of a chemical dimerization drug, rimiducid. Administration of rimiducid dimerizes and activates caspase 9 which activates downstream caspases, leading to apoptosis potentially within minutes to hours (Di Stasi 2011, Tey 2007).

The gamma retrovirus, SFG.iCaspase9.2ADeltaCD19 (BPZ-1001), consists of inducible caspase 9 (iCasp9) linked, via a 2A-like sequence, to truncated human CD19 (DeltaCD19). The iCasp9 genetic modification, unlike the Herpes Simplex Virus (HSV)-TK based safety gene, is human derived and therefore likely to be less immunogenic. Moreover, pre-clinical and clinical studies show that killing occurs with much greater rapidity (within 3 hours) than with HSV-TK. Further advantages of the iCasp9 system are that killing induced by the dimerizer drug is primarily restricted to activated/proliferating cells, thus targeting donor alloreactive T cells active in GVHD, but sparing anti-viral donor T cells and potentially anti-tumor specific T cells. Additionally, administration of the commonly used drug, ganciclovir, is not precluded.

# 4.1.2 Rimiducid Dimerizer Drug

Rimiducid is a member of a new class of lipid-permeable compounds termed activating, or dimerizer, drugs that act by inducing clustering of engineered proteins inside cells.


Rimiducid -inducible activation of the Caspase 9 safety gene is achieved by expressing a chimeric protein (iCasp9), fused to a drug-binding domain derived from human FK506-binding protein (FKBP). This chimeric protein is quiescent inside cells until administration of rimiducid, which cross-links the FKBP domains, initiating iCasp9 signaling. This signaling induces apoptosis of the gene modified cells. Rimiducid is formulated at

#### 4.1.3 CASPALLO Trial

In a Phase I study, ten patients between the ages of 3 and 17 years who had undergone stem-cell transplantation for relapsed acute leukemia were treated with the genetically modified T cells. The cells were detected in peripheral blood and increased in number over time, despite their constitutive transgene expression. A single dose of dimerizing drug, rimiducid, given to the patients in whom GVHD developed, eliminated more than 90% of the modified T cells within 30 minutes after administration and a greater than 90% reduction in CD19+ (i.e. transduced) T cells within 30 minutes of drug administration, and a further log reduction within 24 hours without any reports of infusion toxicity. Moreover, acute GVHD of the skin in all three patients, and of the liver disease in one patient, completely resolved after 24 hours. (Di Stasi 2011). The patients who developed GVHD received rimiducid. None of the 10 patients developed cGvHD. Six of the 10 patients are alive to date, with relapse as the primary cause of death in the other 4 patients (Zhou 2014).

The residual iCasp9 gene modified T cell population expanded over the next 4-14 days and continued to help repopulate the patients' immune systems. The transduced cells were further shown to contain virus and fungal-peptide specific precursor cells which had not caused further GVHD. When examined ex vivo, these non-alloreactive iCasp9 T cells remained susceptible to apoptosis following exposure to the dimerizer rimiducid. The authors concluded that a single dose of dimerizer drug could eliminate the subpopulation of T cells causing GVHD but could spare viral specific cytotoxic T lymphocytes (CTL)s.

The iCasp9 gene is most highly expressed in activated and proliferating T cells, such as those causing GVHD. If cells are not activated, due to lack of viral stimulation for example, expression of the transgene is lower and in a minority of these cells, iCasp9 levels are insufficient to induce apoptosis after single rimiducid dose exposure, allowing subsequent re-expansion (Berger 2004). This hypothesis was supported by the CASPALLO clinical data showing activation-dependent


induction of iCasp9 in T lymphocytes and enhanced susceptibility to dimerizer drug in activated versus resting T cells.

#### 4.2 Evaluation of Benefits/Risks

The direct benefit for the patient will be to improve his clinical outcome in terms of successful eradication of disease, modulation of GVHD and speed of both hematopoietic and immune recovery.

The benefit for the community will be to potentially improve the clinical outcome of patients receiving a HLA-haplo-identical HSCT for the treatment of hematological disorders in terms of: promoting engraftment, lowering TRM and reducing the risk of disease recurrence, thus rendering the procedure more widely applicable.

The potential long term risk of gene therapy using a retroviral vector (although considered a rare risk) is the generation of replication competent retrovirus. While the vector has been constructed to minimize the risk of Replication Competent Retrovirus (RCR), which is therefore considered low risk and unlikely, the inclusion of the safety gene switch and potential to administer rimiducid to rapidly clear the product is a clear advantage of therapy.

# 5 OBJECTIVES OF THE STUDY

# 5.1 Primary Objective

Overall Survival and incidence of Disease-Free Survival in both malignant and non-malignant patients at 1 and 2 years post-transplant. Relapse-Free Survival in malignant patients at 1 year and 2 years post-transplant.

# 5.2 Secondary Objectives

- Long-term survival and safety for a total of 15 years from BPX-501 administration.
- Assessment of PK (rimiducid) and PD (BPX-501) profiles after treatment with rimiducid for aGVHD.

# 5.3 Estimated Enrollment

Up to 175 patients who were previously treated on the BP-004 protocol.

# 5.4 Subject Inclusion Criteria

 Signed written informed consent by the patient or the patient's guardian for children who are minors.


Enrolled on BP-004 protocol, received BPX-501 infusion, completed or discontinued from the study, and are beyond Day +180.

# 5.5 Subject Exclusion Criteria

- Lack of parents'/guardian's informed consent for children who are minors
- Withdrawal from BP-004 study prior to BPX-501 infusion

# 6 PATIENT POPULATION AND SELECTION

This study will enroll any infant (1 day - 23 months), child (2-11 years) or teenager (12-18 years) with malignant hematological disorders in complete morphological remission or non-malignant hematological disorders who did not have a HLA-matched sibling donor and was enrolled on BP-004 and received BPX-501 infusion. No patients between the age of 0-27 days are likely to be enrolled.

#### 6.1 Patient Discontinuation/Withdrawal Criteria

Patients and/or parent(s) or legal guardian(s) are free to discontinue participation or withdraw consent from the long term follow up study at any time, for any reason, and without prejudice to further treatment.

They may withdraw consent to future treatment with rimiducid, or from continuing participation in the LTFU. Patients with difficulty attending visits may stay on study, attend LTFU visits as they are able and remain eligible for rimiducid if needed.

Where possible patients will be encouraged to remain on-study and complete appropriate followup assessments.

If an adverse event (AE) is the reason the patient's treatment is being discontinued by the investigator or the reason that a patient chooses to discontinue treatment, then that adverse event must be documented as the reason for treatment discontinuation.

Patients who discontinue/withdraw from the study will receive treatment as deemed appropriate by their treating physician.

A patient's participation in the study also may be discontinued at any time at the discretion of the investigator. The following may be justifiable reasons for the investigator to remove a patient from the study:

The patient was erroneously included in the long term follow up study.


Data of patients withdrawn from the study will be collected, stored and, whenever indicated, analyzed. These patients will be monitored in terms of outcome with particular regard to survival and, in case of malignancies, risk of recurrence.

If a patient is withdrawn from the study, the investigator should make reasonable effort to complete and report the observations as thoroughly as possible up to the date of withdrawal. All information should be reported on the appropriate case report forms. Data of patients withdrawn from the study will be evaluated, as detailed in the fully executed original consent signed by the patient/parent/guardian upon study entry, unless otherwise indicated. Where possible, these patients will be monitored in terms of outcome for survival and risk of recurrence. The patient/parent/guardian will be informed that follow-up testing or end of study procedures may be required to ensure patient safety is properly maintained.

Patients who have disease relapse or progression should continue to be followed on study to assess survival status and participate in long-term gene therapy monitoring, as appropriate.

Patients that cannot be contacted and who do not have a known reason for discontinuation will be classified as "lost to follow-up" with respect to the reason for discontinuation. The investigator's study staff should make three documented attempts to contact the patient by telephone. If the patient cannot be reached by telephone, the investigator's staff should attempt to contact the patient by certified mail or an alternative similar method, where appropriate.

# 7 DESIGN AND CONDUCT OF THE STUDY

#### 7.1 Trial Rationale

This is a long-term follow-up study evaluating the safety of BPX-501 T cells infused after partially matched, related, T cell-depleted HSCT in pediatric patients previously enrolled on the BP-004 protocol who received BPX-501, completed or discontinued from the study and are beyond Day 180. The trial will evaluate the treatment of GvHD by the infusion of dimerizer drug (rimiducid) in those patients who present with cGvHD who progress or do not respond to standard of care treatment.


# 7.2 Trial Design

The BP-004 Phase I trial design consisted of 3 different escalating doses (2.5x10<sup>5</sup>, 5x10<sup>5</sup>, 1x10<sup>6</sup> cells/kg recipient total body weight) in all patient populations and further escalation of 2 doses (2x10<sup>6</sup>, 4x10<sup>6</sup> cells/kg recipient total body weight) were evaluated in patients with malignant disease only.

Patients were enrolled at the recommended dose for a maximum of 175 pediatric patients total (for both phases), and the minimum active study follow-up for each patient was 180 days in protocol BP-004.

Patients enrolled on the BP-004 study who received BPX-501 T-cells and are beyond Day 180 will be requested to enroll on this long-term follow up protocol, regardless of whether they completed or discontinued from the parent study BP-004.

The follow-up time for evaluation for overall survival and disease-free survival in patients with malignant disease and patients with non-malignant disease will be 1 and 2-years post-transplant. Relapse-free survival in malignant patients will be evaluated at 1 and 2 years. Long term follow-up for survival and gene therapy safety will be 15 years after BPX-501 treatment.

# 7.3 Patient Enrollment, Registration and Assignment to Treatment

Informed consent will be obtained from each patient and/or parent or guardian after the nature of the study is explained and prior to the performance of any study-specific procedures.

Upon enrollment into the study, the patient will continue with the same number assignment as assigned in BP-004.

# 7.4 Rimiducid Dimerizer Drug Packaging, Labeling and Storage

# 7.4.1 Packaging and Formulation

The Rimiducid for Injection is packaged in Type 1 clear glass serum vials (each 3 mL vial contains approximately 2 mL of drug product solution). The contents of each vial is composed

. Each

1476

vial is stoppered with a Teflon® coated serum stopper and a flip-off seal.


# 7.4.2 Labeling

The primary product label (applied directly to the vial) will contain all information for regional use, following the requirements of each competent authority and applicable national and international regulations as described in the pharmacy manual.

# 7.4.3 Storage

The rimiducid for Injection vials must be stored at  $5^{\circ}\text{C} \pm 3^{\circ}\text{C}$  ( $41^{\circ}\text{F} \pm 5^{\circ}\text{F}$ ) in a limited access, qualified refrigerator, preferably without light.

# 7.4.4 Preparation for Treatment

For use, the rimiducid will be diluted prior to administration. The rimiducid is administered via intravenous (IV) infusion at a dose of 0.4 mg/kg diluted in normal saline with volume as appropriate for age of patient to be administered over 2 hours, using a DEHP-free saline bag and solution set.

#### 7.5 Infusion of Rimiducid

# 7.5.1 Chronic GVHD Treatment

Chronic GVHD (cGVHD) typically occurs 100 days or later after HSCT. cGVHD can often present with a sicca-like syndrome with thickened skin, lichen planus, papules, cholestatic jaundice, scleroderma-like skin, eye and GI lesions. cGVHD patients can also develop obstructive pulmonary disease symptoms.

cGVHD is typically classified into mild (i.e., localized skin involvement, with/or without liver dysfunction) or moderate to severe (i.e., generalized skin involvement or localized skin and/or hepatic dysfunction, plus liver histology showing hepatitis/necrosis/cirrhosis, eye involvement, salivary gland involvement, or effects on other organs). Moderate to severe cGVHD usually involves more than one organ with an organ severity score of moderate or greater (or mild or greater for lungs). Management guidelines for cGVHD are shown in Appendix B.

Response should be assessed per Appendix B. Three general categories of overall response are used in clinical trials: complete response (CR), partial response (PR), and lack of response (unchanged, mixed response, progression). Complete response is defined as resolution of all manifestations in each organ or site, and partial response is defined as improvement in at least 1 organ or site without progression in any other organ or site. The 2014 NIH Consensus Working Group recommends that skin, mouth, liver, upper and lower GI, esophagus, lung, eye, and


joint/fascia be considered in evaluating overall response. Genital tract and other manifestations are not included due to lack of validated response measures.

Partial response in a specific organ requires an improvement of 1 or more points on a 4 to 7-point scale or an improvement of 2 or more points on a 10 to 12-point scale. The overall category of PR requires the absence of progression in any organ.

# 7.5.2 Contraception after Rimiducid Infusion

Patients with child-bearing potential (defined as age  $\geq 13$  years) must either commit to true abstinence from heterosexual contact or agree to use and be able to comply with two-physician approved effective contraception methods for 6 months after the last dose of rimiducid.

# 7.6 Monitoring

#### 7.6.1 Rimiducid Response Monitoring

Vital signs are recorded prior to rimiducid infusion, and at 15, 30, 60, 120 and 240 minutes (+/- 5 minutes) after start of infusion. Prior to and after administration of rimiducid, research samples should be collected for BPX-501 T cell tracking and PK testing. Samples for PK testing will be processed differently (Appendix F).

As achievable, and carefully considering patient weight, blood samples should be drawn within 4 hours prior to the initiation of rimiducid infusion; 30 mins after initiation of the infusion; at 2 hours (< 5 min prior to end of the rimiducid infusion), 4 hours, 6 hours, 8 hours, 12 hours, and 24 hours after the initiation of the infusion. Each sample collected out to 24 hours should be split for separate processing. Approximately 0.5 to 1 mL of blood should be processed to plasma and stored at 80° C for later PK analysis of rimiducid. The remaining sample, at least 0.3 mL of blood, should analyzed locally for prompt CD3+CD19+ T cell analysis. Additional samples, at least 0.3 mL, should be drawn at 48 hours and 7 days (after initiation of infusion of each dose of rimiducid), and then at 14 days, 21 days and 28 days after the final dose of rimiducid, in the event multiple doses are administered, for evaluation of T cell responses only.

# 7.6.2 Gene Therapy Monitoring

Long-term follow-up is conducted according to FDA and EMA guidelines Before HSCT and for up to 5-years post stem cell transplant, patients will be evaluated with a physical exam and blood testing testing as outlined below (see Table 2) for vector copy number (VCN) and replication competent retrovirus (RCR) every six months. After 5 years, blood samples will be drawn


annually until 15 years after the last BPX-501 administration. Bellicum will inform the site if sample collection can stop for any patient (criteria for this include all post-treatment PCR assays negative for RCR during the first year, and vector no longer present in 2 consecutive results).

Table 2: Gene Therapy Monitoring Schedule

| Collection Time Point | Clinical Evaluation | Blood (8 mL) |
|---|---|---|
| 1 year | X | X |
| 18, 24, 30, 36, 42, 48, 54, 60 months | X | X* |
| Annually from 6 years to 15 years after the last BPX-<br>501 administration | X | X* |

<sup>\*</sup> Bellicum will inform the site if sample collection can stop for any patient (criteria for this include all post-treatment PCR assays negative for RCR during the first year, and vector no longer present in 2 consecutive results).

# 7.7 Management of Experimental Drugs

Rimiducid will be infused upon the development of GVHD (per instructions in Section 7.2).

This protocol will be conducted during the routine clinical care of the patients. All treatments such as critical medications defined as below shall be collected in the EDC database:

- Treatment for GvHD
- Prophylaxis and/or treatment for infectious complications
- Treatments in association with SAEs

Standard supportive care treatments, non-prescription medications/OTCs, NSAIDs, laxatives/stool softeners, vitamins, and herbal supplements will not be collected if they are not protocol-mandated. Anti-viral prophylaxis will be administered per standard site procedures.

Any post-transplantation pharmacological treatment (including steroids, calcineurin inhibitors, Mycophenolate Mofetil (MMF), Methotrexate (MTX), serotherapy) aimed at preventing GVHD will not be allowed unless approved by Medical Monitor/Sponsor.

# 8 TREATMENTS IN ASSOCIATION WITH SAES EVALUATION CRITERIA

#### 8.1 Laboratory Investigations

Lab tests will be performed according to standard institutional procedures. Additional tests will be undertaken as is the standard institutional practice post-transplant.


# 9 RESPONSE AND TOXICITY EVALUATION

# 9.1 Parameters of safety, assessment of AE and SAE during the duration of the study

# 9.1.1 Safety Parameters and Definitions

Safety assessments will consist of monitoring and recording protocol-defined AEs and SAEs including measurement of protocol-specified hematology, clinical chemistry variables vital signs and other protocol-specified tests that are deemed critical to the safety evaluation of the study drug(s).

The AE grading (severity) scale found in the NCI CTCAE v4.03 will be used for AE reporting. The NCI CTCAE v4.03 can be found:

http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm#ctc 40.

Bellicum or its designee is responsible for reporting relevant SAEs to the FDA other applicable regulatory authorities and participating investigators in accordance with International Conference on Harmonization (ICH) guidelines, FDA regulations, European Clinical Trials Directive (Directive 2001/20/EC) and/or local regulatory requirements.

#### 9.1.2 Adverse Event

An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product or other protocol-imposed intervention, regardless of attribution.

This includes the following:

- AEs not previously observed in the subject that emerge during the protocol specified AE
  reporting period, including signs or symptoms that were not present prior to the AE
  reporting -period.
- Pre-existing medical conditions judged by the investigator to have worsened in severity or frequency or changed in character during the protocol-specified AE reporting period.

#### 9.1.3 Serious Adverse Event

An SAE is any AE that is any of the following:

- Fatal (i.e., the AE actually causes or leads to death)
- Life threatening (i.e.,the AE, in the view of the investigator, places the subject at immediate risk of death)


- Requires or prolongs inpatient hospitalization
- Results in persistent or significant disability/incapacity (i.e., the AE results in substantial disruption of the subject's ability to conduct normal life functions)
- A congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product(s)
- Considered a significant medical event by the investigator (e.g., may jeopardize the subject or may require medical/surgical intervention to prevent one of the outcomes listed above)
- 7. Suspected transmission of infectious agent via a medicinal product

All AEs that meet any of these criteria must be recorded as SAEs, including events that are a normal part of the underlying disease or associated with the general medical management of the patient.

All AEs that do not meet any of the criteria for serious should be regarded as **non-serious AEs**.

The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an AE (as in mild, moderate, or severe pain); the event itself may be of relatively minor medical significance (such as severe headache). "Serious" is a regulatory definition and is based on subject or event outcome or action criteria usually associated with events that pose a threat to a subject's life or vital functions. Seriousness (not severity) serves as the guide for defining regulatory reporting obligations.

Severity and seriousness should be independently assessed when recording SAEs on the electronic Case Report Form (eCRF).

The investigator is responsible for ensuring that all SAEs (as defined in Section 7.1) are recorded on the eCRF and reported to the Sponsor in accordance with protocol instructions.

# 9.1.4 Adverse Event Reporting Period

After informed consent, all adverse events will be reported as per Table 3 which details the guidance for AE reporting after study treatment has initiated.

Table 3: Guidance for Adverse Event Reporting

| Event Type | Reporting Period | Additional Requirements |
|---|---|---|
| OVIID | All cases of GvHD should be reported regardless of onset date and should | Not applicable |


| | not be limited to the below AE/SAE reporting period | |
|---|---|---|
| AEs (post-IMP) | <ul> <li>From the date of BPX-501 infusion until 30 days after administration regardless of causality assessment (including later worsening of events that began during this timeframe).</li> <li>From the date of rimiducid infusion until 30 days after administration regardless of causality assessment.</li> </ul> | Report new AEs for<br>up to 15 years if<br>assessed as related to<br>the investigational<br>products BPX-501<br>and/or rimiducid. |
| SAEs (post-IMP)<br>including Adverse<br>Events of Special<br>Interest* | From the date of BPX-501 infusion until 180 days after administration regardless of causality assessment (including later worsening of events that began during this timeframe). From the date of rimiducid infusion until 30 days after administration regardless of causality assessment. | <ul> <li>Report new SAEs for up to 15 years if assessed as related to the investigational products BPX-501 and/or rimiducid.</li> <li>Report diagnosis of any new secondary malignancy regardless of relationship to investigational product for up to 15 years.</li> </ul> |
| Pregnancy of patients or partner | 12 months after administration<br>of BPX-501 or rimiducid,<br>whichever occurs later. | Report diagnosis of<br>any congenital<br>anomaly in offspring<br>from a study<br>participant or partner<br>for up to 15 years. |

<sup>\*</sup> Adverse Events of Special Interest are Grade III-V encephalopathy or neurologic events - these should be reported to the Sponsor expeditiously, irrespective of regulatory seriousness criteria.

# 9.1.5 GVHD Adverse Event Reporting

All occurrences of GVHD will be reported as Adverse Events (or SAEs) regardless of their start date in relation to study treatment. GVHD events will also be followed until resolution and not limited to the standard AE/SAE reporting period.


# 9.2 Expedited Reporting Requirements for Serious Adverse Events

# 9.2.1 Reporting Requirements for Fatal/Life-Threatening SAEs Related to Investigational Product

Any life-threatening or fatal SAE that is attributed by the investigators to the investigational product will be telephoned to the Medical Monitor immediately, followed by submission of written case details on a CRF within 24 hours.

Sponsor Primary Medical Contact

| Contact | Melissa Aldinger |
|---|---|
| Email | maldinger@bellicum.com |
| Telephone No. | 1-415-656-6341 |
| Contact for SAE Reporting | FAX No.: 617-315-4825/ +34-976 20 44 02 (EU)<br>E-Mail: BellicumSafety@pharmalex.com |

#### Medical Monitor

| Medical Monitor | Swati Gupta Karia, MD,<br>PharSafer Associates Ltd, |
|-----------------|-----------------------------------------------------|
| | White Hart Meadows, Ripley, Surrey GU23 6ND, UK |
| Email | swatigupta@pharsafer.com |
| Telephone No. | Mobile: +44 (0) 7576575575 |

# 9.2.2 Reporting SAEs to the IRB or Ethics Committee and Regulatory Authorities

The investigator must comply with the applicable regulatory requirements related to the reporting of SAEs to the required ECs or IRBs.

All events qualifying as Suspected Unexpected Serious Adverse Reactions (SUSARs) will be reported to the relevant regulatory authorities, central Ethics Committees and to EudraVigilance by the Sponsor or its representative. SUSARs are required to be reported within 7 calendar days for life threatening events and those resulting in death, or 15 calendar days for all others. These timeframes begin with the first notification of the SUSAR to the Sponsor from the investigator.

# 9.2.3 Special Reporting Requirements for Neurotoxicity

BPX-501 cells have been documented to enter the CNS. As the significance of this finding is unknown, all CNS events with apparent encephalitis of ≥ Grade 3 severity must be reported to Bellicum- within the 24 hours (SAE reporting timelines).

Refer to Appendix E for guidelines pertaining to monitoring and management of neurotoxicity.


Record all case details that can be gathered within the reporting timeframe (24 hours) on the Bellicum SAE Report Form and submit the report to re

Guidelines for medical management of neurotoxicity are provided in Appendix E.

# 9.2.4 Reporting Requirements for All SAEs

All SAEs must be reported to Bellicum (via Pharmalex) within 24 hours of learning of the event using the Bellicum SAE Report Form.

For initial SAE reports, investigators should record all case details that can be gathered within the reporting timeframe (24 hours) on the Pharmalex SAE Report Form and submit the report to Follow-up information should be collected on the Pharmalex SAE Report Form as soon as it becomes available.

If local laws require that the site submit all SAEs then the local law will supersede the protocol requirements.

# 9.2.5 Type and Duration of Follow-Up of Patients after Adverse Events

The investigator should follow all unresolved AEs and SAEs until the events are resolved or stabilized, the subject is lost to follow up, or it has been determined that the study treatment or participation is not the cause of the AE/SAE. Resolution of AEs and SAEs (with dates) should be documented on the AE Case Report Form (CRF) or eCRF and in the subject's medical record to facilitate source data verification.

For some SAEs, the Sponsor or its designee may follow up with the site by telephone, fax, electronic mail, and/or a monitoring visit to obtain additional case details deemed necessary to appropriately evaluate the SAE report (e.g., hospital discharge summary, consultant report, or autopsy report).

# 9.2.6 Post-Study Adverse Events

The investigator should notify the study Sponsor of any death or other SAE occurring at any time after a subject has discontinued or terminated study participation if felt to be related to prior study treatment. The Sponsor should also be notified if the investigator should become aware of the development of cancer or of a congenital anomaly in a subsequently conceived offspring of a


subject that participated in this study. The investigator should report these events to Bellicum on the study CRF or eCRF. If the study CRF of eCRF system is no longer available, the investigator should report the event directly to Bellicum via phone or email

# 9.3 End of Study

The study will evaluate overall survival and disease-free survival for all patients enrolled at 1 and 2 years post-transplant. Patients will be followed for a total of 15 years after BPX-501 treatment for gene therapy safety events. The study will be closed after the completion of the 15 years of follow-up.

# 10 DATA COLLECTION, QUALITY ASSURANCE AND MANAGEMENT

# 10.1 Recording of Data

Data will be recorded on an electronic database and will be entered after validation into a computer system for subsequent tabulation and analyses. The investigator must ensure that each subject's anonymity is maintained. Patients will be identified by a unique subject identification number. Study related documents should be kept in strict confidence by the investigator in compliance with applicable regulations and ICH Good Clinical Practice (GCP) Guidelines.

# 10.2 Data Quality Assurance

The investigators undertake to perform the study in accordance with this protocol, GCP and the applicable regulatory requirements.

The investigators are required to ensure compliance with the investigational product schedule, visits schedule and procedures required by the protocol.

The investigators agree to provide all information requested in the Case Report Form in an accurate and legible manner.

# 10.3 Data Management

The investigator will fill in eCRF for documentation. All relevant data collected during the study for all of the patients enrolled into the study have to be entered into the database by the responsible investigator or someone authorized by him/her in a timely manner. The principal investigator (PI) will review all the eCRFs of each patient and confirm the completeness, medical correctness and plausibility of the documented data by signing on all eCRF pages.


Additions and corrections in the eCRF will be dated and signed by the responsible investigator or an authorized person. Reasons must be given for corrections that are not self-explanatory.

Bellicum or the Contract Research Organization (CRO) will ensure that the clinical trial is conducted, recorded, and reported in accordance with the protocol, ICH-GCP, and the applicable regulatory requirement(s).

Representatives of Bellicum or the CRO must be allowed to visit all study site locations periodically to assess the data, quality and study integrity. On-site they will review study records and directly compare them with source documents and discuss the conduct of the study with the investigator, and verify that the facilities remain acceptable. Source documents are defined as: patient files, letters, and laboratory/histology records.

#### 10.4 Statistical Methods

# 10.4.1 Sample Size Determination

The sample size is identical to BP-004 as it is the long term follow-up of those patients.

# 10.4.2 General Statistical Approach

Descriptive statistics will be utilized to summarize overall survival, RFS, DFS, GvHD rates, clinical and biologic response and other measures of safety and toxicity in those patients who received rimiducid administration as well as for the whole population. The analysis population will be stratified by malignant and non-malignant indications.

Data per cohort will be presented, stratified according to the type of disorder, e.g. malignant or non-malignant.

All summary tables for quantitative parameters will display mean, standard deviation, median, range (minimum and maximum), as well as number of missing data, where relevant. All summary tables for qualitative parameters will display counts, percentages, and, number of missing data, where relevant.

# 10.4.3 Study Patient Description

# 10.4.3.1 Disposition of Patients

The number of enrolled patients will be summarized by country, center, and dose using counts and percentages.


# 10.4.4 Demographic and Baseline Characteristics

Baseline characteristics will be described using the patient populations and their accompanying donors. Demographics, medical history, qualifying disorder, and other baseline variables will be summarized as appropriate to the type of data.

# 10.4.5 Endpoint Analysis

# 10.4.5.1 Analysis of Overall Survival

Overall survival, measured as the period of time from the start of the treatment that the patients are still alive at 1 year and 2 years post-transplant will be assessed and reported.

# 10.4.5.2 Analysis of Graft Failure

Secondary graft failure is defined as initial neutrophil engraftment followed by subsequent decline in neutrophil counts  $< 500 \text{ cells/}\mu\text{L}$ , unresponsive to growth factor therapy.

# 10.4.5.3 Analysis Chronic GVHD

The time and severity of cGVHD are graded according to NIH Consensus Criteria (Appendix A).

The initial incidence of severe cGVHD at 6 months will be determined for and will be analyzed by conditioning regimen, αβ T cell dose, disease status, and degree of HLA match. The response rates of cGVHD in patients receiving rimiducid treatment will be determined at 6 months and analyzed by the number rimiducid infusion and time to resolution of cGVHD after rimiducid infusion.

# 10.4.5.4 Analysis of Time to Disease Relapse

To assess the incidence of acute leukemia relapse from the day of transplant, a cumulative incidence curve will computed along with a 95% confidence interval. Death prior to relapse will be considered a competing risk.

# 10.4.5.5 Transplant-Related Mortality

The follow-on protocol will determine long-term TRM/Non-Relapse Mortality at 1 year and 2 years, followed by safety evaluations for gene therapy for 15 years.

#### 10.4.5.6 Immune Reconstitution

Kinetics representing measurements over time within a patient will be generated to visualize general patterns of immune reconstitution. The proportion of iCasp9 positive cells will also be


summarized at each time point. We will also evaluate any indication of differences immune reconstitution across different disease populations.

#### 10.4.6 Safety Analysis

Safety analysis will investigate the analysis populations over the time period defined as from the infusion date of the respective treatment to study end date.

# 10.4.6.1 Adverse Events (AEs)

All adverse events recorded during the study will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) and be graded according to the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) v4.03 scale (see Appendix D).

AEs will be summarized for the following:

- Number (%) of patients with any AE,
- Number (%) of patients with any SAE,
- Number (%) of patients permanently withdrawn from study due to an AE.

All summaries will be presented by treatment group and stratified by type of disorder (e.g. malignant or non-malignant). They will include overall frequency of patients with events as well as frequency of patients with events by primary system organ class and preferred term. A patient will only be counted once within each system organ class and preferred term. For summaries regarding severe or study-drug related AEs, the highest severity or relationship will be considered for each patient per preferred term.

# 10.4.6.2 Deaths, SAEs, and AEs Leading to Treatment Discontinuation

SAEs, events leading to death, and AEs leading to treatment discontinuation will be summarized overall as well as by primary system organ class and preferred term.

# 10.5 Reporting of Deviations to the Protocol

All the deviations to the protocol will be described and justified in a separate form.

# 11 ETHICAL ISSUES/CONSIDERATIONS

#### 11.1 Institutional and Ethical Review

The study will be conducted according to the ethical principles of the declaration of Helsinki, the ICH-GCP Guidelines, the EU Clinical Trial Directive (2001/120/EG), Italian Ministry of Health


(decree of July 15, 1997), Saudi Food and Drug Authority, FDA and other international regulatory agencies.

# 11.2 Investigator's Responsibilities

Any investigator or co-investigator who signed this protocol agrees to carry out this research in accordance with the protocol approved by the ethical committee, GCP and regulatory requirements. Study personnel involved in conducting this trial will be qualified by education, training, and experience to perform their respective task(s). The PI has the right to prematurely discontinue the study for significant efficacy or safety problems and will notify the co-investigators in writing, as well as the ethics committees and the competent authorities according to law and regulations.

#### 11.2.1 Patient Informed Consent

The patient or parents/legal guardians are to be informed both in writing and verbally by the investigating physician. The patient and his/her parents/guardians must be given ample opportunity to decide whether or not to participate in this study and to ask questions concerning this. It must also be made clear to the patient that he/she can withdraw from the study at any time without giving reasons and that he/she will not be in any way disadvantaged by this. Assent will be documented as required by the IRB or the EC. The informing physician, the patient or guardian must each personally date and sign an informed consent form with a declaration on data privacy. Any informed consent will be part of the investigator's file and retained with it. The patient will retain a copy of the patient information.

#### 11.2.2 Data Management and Storage

The investigator will organize the storage of the identification codes of the patients for at least 15 years after the end of the study. The files of the patients (medical records) and other original data will be kept for a minimum period of 15 years. Relevant parts of those records specific to support the traceability of BPX-501 from donor to recipient will be retained as applicable by the investigator, manufacturer and Sponsor per local requirement.


# 12 REFERENCES

Amrolia PJ, Muccioli-Casadei G, Huls H, et al. Adoptive immunotherapy with allodepleted donor T-cells improves immune reconstitution after haploidentical stem cell transplantation. *Blood*. 2006; 108:1797-1808.

Berger C, Blau C A, et al. Pharmacologically regulated Fas-mediated death of adoptively transferred T cells in a nonhuman primate model. *Blood*. 2004; 103:1261-1269.

de Brabander C, et al. Increased incidence of neurological complications in patients receiving an allogeneic bone marrow transplantation from alternative donors. J Neurol Neurosurg Psychiatry. 2000,68:36-40.

Di Stasi A, Tey S-K, Dotti, G et al. Inducible Apoptosis as a Safety Switch for Adoptive Cell Therapy. N Engl J Med. 2011; 365:1673-83.

Dowling MR, Li S, Dey BR, SL McAfee, et al. Neurologic complications after allogeneic hematopoietic stem cell transplantation: risk factors and impact *BMT*. 2018; 53:199-206.

Engelborghs S, et al. Consensus guidelines for lumbar puncture in patients with neurological diseases. *Elsevier*. 2017;8:111-126.

Folstein MF, et al. "Mini-mental state": a practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res 1975:12:189-198.

Rocha V, Locatelli F. Searching for alternative donors of haematopoietic stem cell for paediatric patients. *Bone Marrow Transplant*. 2008; 41:207-214.

Syed FI, et al. Central nervous system complications of hematopoietic stem cell transplant. Hematol Oncol Clin N Am 2016;30:887-898.

Tey SK, Dotti G, Rooney CM, et al. Inducible caspase 9 suicide gene to improve the safety of allodepleted T cells after haploidentical stem cell transplantation. *Biol Blood Marrow Transplant*. 2007: 13:913-24.

Uckan D, et al. Life-threatening neurological complications after bone marrow transplantation. Bone Marrow Transplant 2005, 35:71-76.

Zhou X, Di Stasi A, Tey SK, et al. Long-term outcome after haploidentical stem cell transplant and infusion of T cells expressing the inducible caspase 9 safety transgene. *Blood*. 2014;123(25):3895-3905.


# Appendix A: Chronic GVHD Grading Scale and Assessment Appendix A.1: NIH Consensus Grading Chronic GVHD

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| PERFORMANCE<br>SCORE:<br>KPS ECOG LPS | ☐ Asymptomatic<br>and fully active<br>(ECOG 0; KPS or<br>LPS 100%) | ☐ Symptomatic,<br>fully ambulatory,<br>restricted only in<br>physically strenuous<br>activity (ECOG 1,<br>KPS or LPS 80-<br>90%) | ☐ Symptomatic,<br>ambulatory,<br>capable of self-<br>care, >50% of<br>waking hours out<br>of bed (ECOG 2,<br>KPS or LPS 60-<br>70%) | Symptomatic,<br>limited self-care,<br>>50% of waking<br>hours in bed (ECOG<br>3-4, KPS or LPS<br><60%) |
| SKIN Clinical features: Maculopapular rash Lichen planus-like features Papulosquamous lesions or ichthyosis Hyperpigmentation Keratosis pilaris Erythema Erythroderma Poikiloderma Sclerotic features Pruritus Hair involvement Nail involvement SBA involved | □ No Symptoms | □ <18% BSA with disease signs but NO sclerotic features | ☐ 19-50% BSA OR involvement with superficial sclerotic features "not hidebound" (able to pinch) | □ >50% BSA OR<br>deep selerotic<br>features "hidebound"<br>(unable to pinch) OR<br>impaired mobility,<br>ulceration or severe<br>pruritus |
| Моитн | □ No symptoms | ☐ Mild symptoms<br>with disease signs<br>but not limiting oral<br>intake significantly | ☐ Moderate<br>symptoms with<br>disease signs with<br>partial limitation of<br>oral intake | Severe symptoms<br>with disease signs on<br>examination with<br>major limitation of<br>oral intake |
| EYES Mean tear test (mm): □ >10 □ 6-10 □ ≤5 □ Not done | □ No symptoms | ☐ Mild dry eye symptoms not affecting ADL (requiring eyedrops ≤ 3 x per day) OR asymptomatic signs of keratoconjunctivitis sicca | ☐ Moderate dry eye symptoms partially affecting ADL (requiring drops > 3 x per day or punctal plugs), WITHOUT vision impairment | ☐ Severe dry eye symptoms significantly affecting ADL (special eyeware to relieve pain) OR unable to work because of ocular symptoms OR loss of vision caused by keratoconjunctivitis sicca |
| GI TRACT | □ No symptoms | ☐ Symptoms such<br>as dysphagia,<br>anorexia, nausea,<br>vomiting, abdominal<br>pain or diarrhea<br>without significant<br>weight loss (<5%) | Symptoms associated with mild to moderate weight loss (5-15%) | Symptoms associated with significant weight loss >15%, requires nutritional supplement for most calorie needs OR esophageal dilation |
| LIVER | □ Normal LFT | ☐ Elevated<br>Bilirubin, AP*, AST<br>or ALT <2 x ULN | ☐ Bilirubin >3<br>mg/dl or Bilirubin,<br>enzymes 2-5 x<br>ULN | ☐ Bilirubin or enzymes > 5 x ULN |


# Appendix A.1 NIH Consensus Grading Chronic GVHD (cont)

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| Lungs' | □ No symptoms | <ul> <li>Mild symptoms<br/>(shortness of breath<br/>after climbing one<br/>flight of steps)</li> </ul> | Moderate<br>symptoms<br>(shortness of<br>breath after<br>walking on flat<br>ground) | Severe symptoms (shortness of breath at rest; requiring 0 <sub>2</sub> ) |
| DLCO | ☐ FEV1 > 80% <b>OR</b><br>LFS=2 | ☐ FEV1 60-79%<br>OR LFS 3-5 | ☐ FEV1 40-59%<br>OR LFS 6-9 | ☐ FEV1 ≤39% <b>OR</b><br>LFS 10-12 |
| OINTS AND<br>PASCIA | □ No symptoms | ☐ Mild tightness of<br>arms or legs, normal<br>or mild decreased<br>range of motion<br>(ROM) AND not<br>affecting ADL | ☐ Tightness of arms or legs OR joint contractures, erythema thought due to fasciitis, moderate decrease ROM AND mild to moderate limitation of ADL | ☐ Contractures WITH significant decrease of ROM AND significant limitation of ADL (unable to tie shoes, button shirts, dress self etc.) |
| | □ No symptoms clinical manifestations of the severity (0-3) based on | | | |
| , severe – 3) | is severity (0-3) based on | its functional impact wi | теге аррисаоте (попе | - 0,mild -1, moderate |
| sophageal strictur | re or web Pericardi | al Effusion | Pleural Effusion(s)_ | |
| Ascites (serositis)_ | Nephroti | c syndrome | Peripheral Neuropath | у |
| M yasthenia Gra | vis Cardiom | yopathy | Eosinophilia > 500µl | |
| olymyositis | Cardiac | conduction defects | Coronary artery invo | lvement |
| Platelets <100,000 | /μl Progress | ive onset | | |
| OTHERS: Specify: | | | | |

# Global scoring of cGVHD

| Number of Organs | Mild cGVHD | Moderate cGVHD | Severe cGVHD |
|------------------|------------|----------------|--------------|
| 1 | Score 1 | Score 2 | Score 3 |
| 2 | Score 1 | Score 2 | Score 3 |
| 3 | | Score 1 | Score 3 |
| Lung involvement | | Score 1 | Score 2 |

Mild cGVHD = 1 or 2 organs involved (except for lung) with maximum score of 1 Moderate cGVHD = lung score of 1 or 3 organs with score of 1 or at least 1 organ with score of 2 Severe cGVHD = lung score of 2 or score of 3 in any organ.

#### Reference:

Filipovitch AH et al. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56.


# Appendix A.2: Response Determination for Chronic GvHD

Response Determination for Chronic GVHD Clinical Trials based on Clinician Assessments

| Organ | Complete Response | Partial Response | Progression |
|---|---|---|---|
| Skin | NIH Skin Score 0 after | Decrease in NIH Skin Score | Increase in NIH Skin Score by 1 or |
| | previous involvement | by 1 or more points | more points, except 0 to 1 |
| Eyes | NIH Eye Score 0 after | Decrease in NIH Eye Score | Increase in NIH Eye Score by 1 or |
| | previous involvement | by 1 or more points | more points, except 0 to 1 |
| Mouth | NIH Modified OMRS 0 after | Decrease in NIH Modified OMRS | Increase in NIH Modified OMRS |
| | previous involvement | of 2 or more points | of 2 or more points |
| Esophagus | NIH Esophagus Score O after | Decrease in NIH Esophagus | Increase in NIH Esophagus Score |
| | previous involvement | Score by 1 or more points | by 1 or more points, except 0 to 1 |
| Upper GI | NIH Upper GI Score 0 after | Decrease in NIH Upper GI | Increase in NIH Upper GI Score |
| | previous involvement | Score by 1 or more points | by 1 or more points, except 0 to 1 |
| Lower GI | NIH Lower GI Score 0 after | Decrease in NIH Lower GI | Increase in NIH Lower GI Score by |
| | previous involvement | Score by 1 or more points | or more points, except from 0 to 1 |
| Liver | Normal ALT, alkaline | Decrease by 50% | Increase by 2 × ULN |
| | phosphatase, and Total | | |
| | bilirubin after previous | | |
| | elevation of 1 or more | | |
| Lungs | - Normal %FEV1 after | - Increase by 10% predicted | - Decrease by 10% predicted |
| | previous involvement | absolute value of %FEV1 | absolute value of %FEV1 |
| | - If PFTs not available, NIH | - If PFTs not available, decrease | - If PFTs not available, increase in |
| | Lung Symptom Score 0 | in NIH Lung Symptom Score | NIH Lung Symptom Score by 1 |
| | after previous involvement | by 1 or more points | or more points, except 0 to 1 |
| loints and fascia | Both NIH Joint and Fascia | Decrease in NIH Joint and Fascia | Increase in NIH Joint and Fascia |
| ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | Score 0 and P-ROM score | Score by 1 or more points or | Score by 1 or more points or |
| | 25 after previous involvement | increase in P-ROM score by 1 | decrease in P-ROM score by 1 |
| | by at least 1 measure | point for any site | point for any site |
| Global | Clinician overall severity score 0 | Clinician overall severity score | Clinician overall severity score |
| | | decreases by 2 or more points | increases by 2 or more points |
| | | on a 0-10 scale | on a 0-10 scale |

ULN indicates upper limit of normal.


# Appendix A.3: Chronic GvHD Activity Assessment - Clinician

| rsphegis or<br>od/mopheg | 0 ns | moden ( Licher- ( | erythema or<br>ate erythema<br><25%)<br>like changes<br><25%)<br>and food or pits<br>and foods or pits<br>and foods or pits | bat not | Seven<br>(4<br>Lichen-<br>(2)<br>Ulcers Im | | 2<br>2<br>3 | Severe cryste (225%) Lichen-like cha (>50%) Severe ulceral (>20%) I mucosal cha | inges<br>lions | 3 6 |
|---|---|---|---|---|---|---|---|---|---|---|
| Nane<br>al symptom<br>isphagla or<br>isphagla or<br>od/mophag | 0 ns | hegie with so | <25%) ria food or pilis rid foods or pilis | dwing the | Ulcers Im | 550%)<br>olving (s20%)<br>Total sco | 3 | (>50%)<br>Bevere ulcerat<br>(>20%) | lions | |
| al symptom<br>raphagla or<br>raphagia or<br>od/mophag | ns<br>r odynoph<br>r od/moph | hegie with so | ria fosa or pilis<br>vid fosas or pili | bat not | Ulcers Im | olving (s20%) Total sco | | Severe ulcerat<br>(>20%) | | 6 |
| isphagila or<br>isphagila or<br>odunophagila<br>i | r adynoph<br>r advnoph | hegia with so | ed foods or pet | bat not | | | re for a | I mucosal cha | inges | |
| isphagila or<br>isphagila or<br>odunophagila<br>i | r adynoph<br>r advnoph | hegia with so | ed foods or pet | bat not | | | | | anges | |
| ermittent an | empriorits, | with some n | n in oral intake<br>eduction is ora | during the | lay of the pa<br>post week<br>wing the pas | st week | | ry day of the sest | | |
| guilf stools<br>oose ar liqui<br>ose or liqui<br>o | during the<br>rid stools,<br>id stools t | te past week<br>, on some da<br>throughout th | ys <u>diving the a</u><br>se day, <u>on aims</u> | ast week<br>st every o | lay of the pa | st week, withou | ut requiri | ng intervention to ; | | correct |
| | | | Single Breath | DLCO (ad) | justed for hem | oglobin) | TLG | | RV | |
| | | mg/dL | ALT | UL | ULN | UV. | Alkaine f | hosphatase<br>UL | ULN | w |
| sked in 2 or 9 | 6 Mins. | | Kamofsky or i | arreky | Platelel Co | int | TotalWB | c | Eosinophi | 5 |
| di<br>di | on<br>Warrhao <u>ga</u><br>Fis<br>ibin Ul<br>mg/di. | on<br>Mamhao <u>ya almosti a</u><br>FYC<br>ibin ULN | on diamhea <u>on aimost eveny day of N</u><br>PYC<br>bin ULN<br>ragist, mglet, | on diamhoo on aimosi avery day of the past week in FVC Single Breath thin ULIN ALT mg/st. mg/st. | on Slamboo on almost every day of the past week, requiring PVC Single Breath DLCO (at thin ULN ALT mg/st. Ut. | on disambee on elmost every day of the past week, requiring intervention. FYC Single Breath DLCO (adjusted for hern thin ULN MISS) and ULN MISS. ULN MISS. ULN MISS. ULN | on distribution on admost every day of the past week, requiring intervention to prevent or so FVC Single Bresti D.CO (asjusted for hemoglotin) thin ULN ALT ULN might. ULL UL. UL. | on disambee on almost every day of the east seek, requiring intervention to exercise or general value FVC Single Breati DLCO (adjusted for hemoglobin) TLG thin ULN ALT ULN Alkaine fingfall might ULN UL UL | on Silambee on almost every day of the east seek, requiring intervention to prevent or govern volume depletion. FVC Single Breatt DLCO (adjusted for hemoglobin) TLC thin ULN ALT ULN Alkaline Phosphakee might. UL. UL. UL. UL. | Blambee on almost every day of the past week, requiring intervention to prevent or cornect volume denietion. FVC Single Breath DLCO (adjusted for hemoglobin) TLC RV sibin ULN ALT ULN Alkeline Phosphakese ULN mg/st. ULL UL. UL. UL. |


# Appendix A.3: Chronic GvHD Activity Assessment - Clinician (cont)

# CHRONIC GVHD ACTIVITY ASSESSMENT- CUNICIAN

| 7 | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| SKIN GVHD features to be scored by BSA: Check all that apply: Maculopapular rash / erythema Lichen planus-like features Sclerotic features Papulosquamous lesions or ichthyosis Keratosis pilaris-like | | □ 1=18% BSA | □ 19-50% BSA | □ >50% BSA |
| Abnormality present but ex | plained entirely by | non-GVHD documente | ed cause (specify): | <u> </u> |
| SKIN FEATURES<br>SCORE: | ☐ No sclerotic features | | ☐ Superficial<br>sclerotic features "not<br>hidebound" (able to<br>pinch) | Check all that apply: Deep selerotic features "Hidebound" (unable to pinch) Impaired mobility Ulceration |
| If skin features score = 3, BS How would you rate the severe and 10 is the most 0 1 2 Symptoms not at all severe | severity of this pati | ent's skin and/or joint t | 9 10<br>Most severe<br>symptoms possible | cale, where 0 is not at all |
| Eyes | ☐ No symptoms<br>symptoms | ☐ Mild dry eye symptoms not affecting ADL (requirement of lubricant eye drops ≤ 3 x per day) | ☐ Moderate dry eye symptoms partially affecting ADL (requiring lubricant eye drops > 3 x per day or punctal plugs), WITHOUT new vision impairment due to KCS | Severe dry eye symptoms significantly affecting ADL (special eyeware to relieve pain) OR unable to work because of ocular symptoms OR loss of vision due to KCS |
| ☐ Abnormality present but ex | plained entirely by | non-GVHD documents | ed cause (specify): | - |
| Lungs | □ No symptoms | ☐ Mild symptoms<br>(shortness of | ☐ Moderate symptoms<br>(shortness of breath | ☐ Severe symptoms<br>(shortness of breath |

## Appendix A.3: Chronic GvHD Activity Assessment - Clinician (cont)

#### CHRONIC GVHD ACTIVITY ASSESSMENT

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| JOINTS AND FASCIA | □ No symptoms | ☐ Mild tightness of<br>arms or legs, normal<br>or mild decreased<br>range of motion<br>(ROM) AND not<br>affecting ADL | ☐ Tightness of arms or<br>legs OR joint contractures,<br>crythema thought due to<br>fasciitis, moderate<br>decrease ROM AND mild<br>to moderate limitation of<br>ADL. | ROM AND significant<br>limitation of ADL |



Abnormality present but explained entirely by non-GVHD cause (specify):


Today's Date \_\_\_\_\_

SUBJECT ID \_\_\_\_\_\_

## Appendix A.3: Chronic GvHD Activity Assessment - Clinician (cont)

CHRONIC GVHD ACTIVITY ASSESSMENT-PATIENT SELF REPORT

| Symptoms | | | | | | | | | | | 307470 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Please rate how severe the following<br>symptoms have been in the <u>last seven</u><br><u>days</u> . Please fill in the circle below from 0<br>(symptom has not been present) to 10 (the | | Not<br>Present | | | | | | | | | As Bad As You<br>Can Imagine | |
| symptom was as bad as<br>could be) for each item. | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Your skin itching at its | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Your skin and/or joint<br>their WORST? | tightening at | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Your mouth sensitivity at its WORST? | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Your genital discomfo<br>(Women – vagina, vulv<br>(Men – penis) | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Eyes | What is your | how sev | vere this s | ymptom | | | _ | | | | | |
| | all severe) to | o 10 (mc | ost severe | 9): | | | 0 1 | 2 3 | 4 5 | 6 7 | 8 9 | 10 |
| Patient Global Rating | \$; | | | | | | | | | | | |
| | nk that your chron | ic graft | versus h | ost disea | se is mi | ld, mode | rate or s | evere? | | | | |

Most severe cGvHD symptoms possible

0 1 2 3 4 5 6 7 8 9 10

3. Compared to a month ago, overall would you say that your cGvHD symptoms are:

+3= Very much better +2= Moderately better +1=A little better

+1=A little better 0= About the same -1=A little worse -2=Moderately worse -3=Very much worse


# Appendix B: Management of Chronic GVHD (cGVHD)

| Event | Management |
|---|---|
| cGVHD - Mild | Consider tissue biopsy to establish diagnosis |
| | Initial treatment with topical or IV steroids, or other systemic treatments (eg, calcineurin inhibitors), per institutional standard of care for mild cGVHD should be instituted. Guidelines for topical corticosteroid treatment include |
| | the following (Couriel 2006): |
| | <ul> <li>Face, axillae, and groin: lower potency steroids (hydrocortisone 1-2.5%, desonide 0.05%)</li> <li>From the neck down: mid-strength steroids (e.g., triamcinolone</li> </ul> |
| | 0.1% cream or ointment) |
| | <ul> <li>Systemic corticosteroids when used should be administered as<br/>methylprednisolone 2 mg/kg/day IV in a single dose; or a dose equivalent of<br/>prednisone or dexamethasone) (Martin 1990; see also corticosteroid</li> </ul> |
| | conversion table C below). |
| | If no response to steroids/systemic therapies occurs within 7 days, or there is a worsening in cGVHD, patients may then receive rimiducid: |
| | <ul> <li>Adults: 40 mg IV</li> <li>If there is evidence of clinical improvement (e.g. partial response) but not complete resolution after the first dose of rimiducid, then rimiducid may be repeated up to a total of 3 doses beginning 48 hours after the first dose, with each dose separated by 48 hours</li> </ul> |
| | <ul> <li>Daily examination on day 1 and day 2 should be performed after initiating treatment with rimiducid, then weekly for 1 month, every 2 weeks for 100 days, and monthly after 100 days post-rimiducid administration</li> <li>For new or recurrent cGVHD episodes, rimiducid may be</li> </ul> |
| | considered for repeat administration with the above guidelines if the investigator considered rimiducid to offer clinical benefit with prior episodes. |
| | <ul> <li>If no response to topical steroids or rimiducid, the investigator should<br/>consider other medications per institutional guidelines (eg, calcineurin<br/>inhibitors, sirolimus, mycophenolate).</li> </ul> |
| | Peripheral blood will be used to evaluate BPX-501 cells (CD3+CD19+) at the following times: Prior to administration of systemic continuously described described. |
| | <ul> <li>Prior to administration of systemic corticosteroid doses (e.g,<br/>methylprednisolone), at 4 and 24 hours (± 30 minutes) post-<br/>systemic corticosteroid doses, and at 7, 14, 21 and 28 days<br/>(± 24 hours) post-systemic corticosteroid doses</li> </ul> |
| | When possible, considering patient weight, blood samples will be drawn within 4 hours (± 30 minutes) prior to the initiation of rimiducid infusion; 30 mins (± 5 minutes) after initiation of the infusion; at 2 hours (< 5 min prior to end of the rimiducid infusion), 4 hours, 6 hours, 8 hours, 12 hours, and 24 hours (± 30 minutes) |
| | after the initiation of the infusion. Each sample collected out to 24 hours should be split for separate processing. Approximately 0.5 to 1 mL of blood should be processed to plasma and stored at -80 C |
| | for later PK analysis of rimiducid. The remaining samples, at least 0.3 mL of blood, should be analyzed locallyfor prompt CD3+CD19+ T cell analysis. These additional samples (at least 0.3 mL) will be drawn at 48 hours (± 30 minutes), then at 7 days (after |
| | initiation of infusion of each dose of rimiducid), and at 14 days, 21 days, and 28 days (± 24 hours) after the final dose of rimiducid (in |


| | the event multiple doses are administered) and evaluated for T cell |
|---|---|
| | responses only. |
| | At each evaluation, complete Chronic GVHD Activity Assessment- |
| | Clinician and Chronic GVHD Activity Assessment-Patient Self Report |
| cGVHD – Moderate | Consider tissue biopsy to establish diagnosis |
| to Severe | <ul> <li>Initial treatment with IV steroids or other systemic treatments (eg,</li> </ul> |
| to severe | calcineurin inhibitors) per institutional standard of care for extensive |
| | cGVHD should be instituted. |
| | If no response to topical steroids or rimiducid, the investigator should |
| | consider other medications per institutional guidelines (eg, calcineurin |
| | inhibitors, sirolimus, mycophenolate). |
| | If no response steroids/systemic therapies occurs within 7 days, or there is a |
| | worsening in cGVHD, patients may then receive rimiducid |
| | o Children: 0.4 mg/kg to a maximum of 40 mg IV |
| | o Adults: 40 mg IV |
| | o If there is evidence of clinical improvement (e.g. partial response) |
| | but not complete resolution after the first dose of rimiducid, then |
| | rimiducid may be repeated up to a total of 3 doses beginning 48 |
| | hours after the first dose, with each dose separated by 48 hours |
| | <ul> <li>Daily examination on day 1 and day 2 should be performed after</li> </ul> |
| | initiating treatment with rimiducid, then weekly for 1 month, every |
| | 2 weeks for 100 days, and monthly after 100 days post-rimiducid |
| | administration |
| | o For new or recurrent cGVHD episodes, rimiducid may be |
| | considered for repeat administration with above guidelines if the investigator considered rimiducid to offer clinical benefit with prior |
| | episodes |
| | <ul> <li>Peripheral blood will be used to evaluate BPX-501 cells (CD3+CD19+) at</li> </ul> |
| | the following times: |
| | Prior to administration of systemic corticosteroid doses (e.g., |
| | methylprednisolone), at 4 hours and 24 hours (± 30 minutes) post- |
| | systemic corticosteroid doses, and at 7, 14, 21 and 28 days (± 24 |
| | hours) post-systemic corticosteroid doses |
| | <ul> <li>As achievable, considering patient weight, blood samples will be</li> </ul> |
| | drawn within 4 hours (± 30 minutes) prior to the initiation of |
| | rimiducid influsion; 30 mins (± 5 minutes) after initiation of the |
| | infusion; at 2 hours (< 5 min prior to end of the rimiducid infusion), |
| | 4 hours, 6 hours, 8 hours, 12 hours, and 24 hours (± 30 minutes) |
| | after the initiation of the infusion. Each sample collected out to 24 |
| | hours should be split for separate processing. Approximately 0.5 to |
| | 1 mL of blood should be processed to plasma and stored at -80 C |
| | for later PK analysis of rimiducid. The remaining samples, at least 0.3 mL of blood, should be analyzed locallyfor prompt |
| | CD3+CD19+ T cell analysis. These additional samples (at least 0.3 |
| | mL) will be drawn at 48 hours (± 30 minutes) and 7 days (± 24 |
| | hours) (after initiation of infusion of each dose of rimiducid), and |
| | then at 14 days, 21 days, and 28 days (± 24 hours) after the final |
| | dose of rimiducid (in the event multiple doses are administered) and |
| | evaluated for T cell responses only. |
| References: | |

#### References:

Couriel D, et al. Ancillary therapy and supportive care of chronic graft-versus-host disease: NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: V. Ancillary Therapy and Supportive Care Working Group Report. Biology of Blood and Marrow Transplant 2006;12:375-396. Martin PJ, et al. A retrospective analysis of therapy for acute graft-versus-host disease: initial treatment. Blood 1990;76:1464-1472.


**Appendix C: Corticosteroid Conversion Table** 

| Cortico | steroid Conversion T | `able |
|--------------------|----------------------------------|----------------|
| Glucocorticoid | Approximate equivalent dose (mg) | Half-life (hr) |
| | Short-Acting | |
| Cortisone | 25 | 8-12 |
| Hydrocortisone | 20 | 8-12 |
| | Intermediate-Acting | |
| Methylprednisolone | 4 | 18-36 |
| Prednisolone | 5 | 18-36 |
| Prednisone | 5 | 18-36 |
| Triamcinolone | 4 | 18-36 |
| | Long-Acting | |
| Betamethasone | 0.6 - 0.75 | 36-54 |
| Dexamethasone | 0.75 | 36-54 |

Dixon JS. Second-line Agents in the Treatment of Rheumatic Diseases. Informa Health Care, 1991. (456). Melkle AlW and Tyler FH. Potency and duration of action of glucocorticoids. Am J of Med 1977;63;200. Webb R, Singer M. Oxford Handbook of Critical Care. Oxford; New York: Oxford University Press, 2005.


## Appendix D: AE Grading and Toxicity

The AE grading (severity) scale found in the NCI CTCAE v4.03 will be used for AE reporting.

The NCI CTCAE v4.03 can be found:

http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm#ctc 40

AE Grading (Severity) Scale

| Grade | Severity | Alternate Description a |
|---|---|---|
| 1 | Mild (apply event-specific<br>NCI CTCAE grading criteria) | Transient or mild discomfort<br>(< 48 hours); no interference<br>with the subject's daily<br>activities; no medical<br>intervention/therapy required |
| 2 | Moderate (apply eventspecific-<br>NCI CTCAE grading criteria) | Mild to moderate interference<br>with the subject's daily<br>activities; no or minimal<br>medical intervention/therapy<br>required |
| 3 | Severe (apply event-specific<br>NCI CTCAE grading criteria) | Considerable interference with<br>the subject's daily activities;<br>medical intervention/therapy<br>required; hospitalization<br>possible |
| 4 | Very severe, life threatening,<br>or disabling (apply eventspecific<br>NCI CTCAE grading criteria-) | Extreme limitation in activity;<br>significant medical<br>intervention/therapy required,<br>hospitalization probable |
| 5 | Death related to AE | |

<sup>&</sup>lt;sup>a</sup>Use these alternative definitions for Grade 1, 2, 3, and 4 events when the observed or reported AE is not in the NCI CTCAE listing.


### Appendix E: Guidelines for Monitoring & Management of Neurotoxicity

Neurologic complications occur in approximately 6.4-19.2% (Dowling 2017, Syed 2016, Uckan 2005) of patients after allogeneic hematopoietic stem cell transplantation. They are the cause of death in 10-15% of children undergoing allogeneic HSCT (Uckan 2005). Children who develop encephalopathy have a poor prognosis, with a minority experiencing partial or complete neurologic recovery. The etiologies of these complications are diverse and include infection, posterior reversible encephalopathy syndrome (PRES), metabolic encephalopathy, medications, GVHD, hemorrhage, multi-organ dysfunction, and inflammatory conditions. Risk factors for these complications include acute GVHD, thrombocytopenia, delayed platelet engraftment, primary underlying disease, and age (Dowling 2017, Syed 2016, Uckan 2005). CNS toxicity may occur at different rates among different donor sources (matched unrelated or haploidentical donors have a higher rate than matched related donors) (de Brabander 2000).

Particular attention should be paid to the onset of Grade 2 or higher level of depressed consciousness, encephalopathy, hypersomnia, lethargy, leukoencephalopathy, meningismus, myelitis, reversible posterior leukoencephalopathy syndrome (PRES), seizure, or somnolence.

Diagnostic evaluation should include assessment of focal versus generalized type of symptoms. Generalized findings may include seizures, metabolic encephalopathy, or infection, while focal findings raise suspicion for mass lesions, hemorrhage, stroke, or spinal cord abnormalities (Syed 2016, Uckan 2005).

Guidelines monitoring of neurotoxicity are provided in Table E.1. Patients should undergo a daily neurologic examination and mini-mental status examination (MMSE) (Folstein 1975) or modified mini mental status examination (pediatric population) while inpatient during the hematopoietic stem cell transplant, both before and after infusion of BPX-501. Some pediatric populations (<3 years old) are exempt from completing this examination Daily neurologic examinations should also be performed during any readmissions after allogeneic HSCT. A neurologic examination should be performed as part of all routine clinical follow-up examinations during each outpatient visit while patients are being treated on BPX-501 clinical trials.

In the event of the development of Grade 2 or higher nervous system or mental status changes, refer to Table E.2 below for evaluation and management guidelines.

In cases where a lumbar punctures (LP) is potentially warranted to evaluate the cerebrospinal fluid (CSF) to aid in the differential diagnosis of clinical neurological changes, procedures and precautions should be taken to rule out contraindications for performing an LP (Table E.3), consistent with consensus guidelines for performing LPs in patients with neurological diseases (Engelborghs 2017).

If a diagnostic LP is performed, attempts should be made to minimize side effects such as infections, pain and post-LP headaches, including, but not limited to: a) use of 25G atraumatic type needles, b) performing 4 or less attempts, c) passive CSF collection instead of active CSF withdrawal using a syringe, d) collection of less than 30 mL of CSF, and e) lateral recumbent position (see Table E.3; Engelborghs 2017).


Table E.1: Monitoring of Patients for Neurologic Complications

| Timing | Neurologic examination | Mini-mental status<br>examination |
|---|---|---|
| Routine outpatient clinic visits<br>or emergency room visits | ✓ | ✓ |
| Change in mental status or<br>presence of CNS dysfunction<br>(e.g., reduced consciousness,<br>delirium) | ~ | ~ |

Version 3.0  1503

Table E.2: Management Guideline for Neurotoxicity\*

| Table E.2: | Management Guideline for Neurotoxicity* |
|---|---|
| Event | Management |
| Grade ≥ 2 (Focal) <sup>1</sup> | <ul> <li>Consider neurology consultation and performing EEG</li> <li>Perform daily neurological and mini-mental status examinations during</li> </ul> |
| | hospitalizations to evaluate for resolution/worsening of symptoms |
| | <ul> <li>Perform CNS imaging (MRI and/or contrast enhanced CT)</li> </ul> |
| | <ul> <li>Consider CSF evaluation for presence of cell counts (and differential),</li> </ul> |
| | glucose, protein and gram-stain for bacteria. |
| | <ul> <li>CSF evaluations for other infectious etiologies (e.g., herpes viruses,</li> </ul> |
| | JC virus, fungal, West Nile virus and toxoplasma) |
| | <ul> <li>CSF samples should be sent to the Sponsor for research use to<br/>evaluate for the presence of BPX-501 cells</li> </ul> |
| | Consider empiric use of anticonvulsants if seizure is expected |
| | Special consideration should be considered for conditioning agents |
| | (e.g., Busulfan) or prophylactic GVHD medications (e.g.,<br>calcineurin inhibitors) as an etiology and institutional guidelines |
| | should be instituted for possible treatments (eg, prophylactic GVHD |
| | medication changes and/or treatment with seizure medications) |
| | Start management of stroke/ischemia per institutional guidelines if suspected |
| | <ul> <li>Administration of antiviral and/or anti-fungal therapy as per institutional</li> </ul> |
| | standard of care should be considered if infectious etiology is suspected |
| | (tailored for lab data results) |
| | A brain biopsy should be considered if other diagnostic tests are unrevealing |
| | as to an etiology. |
| | <ul> <li>Rimiducid may be administered if CNS infection ruled out and no<br/>improvement after 48 hours of high-dose corticosteroids (1000 mg/day x 2</li> </ul> |
| | days for adults or 30 mg/kg/day x 2 days in children) rimiducid may be |
| | administered in conjunction with corticosteroids and anti-infective agents. |
| | Samples for PK analysis of rimiducid for research use, should be collected |
| | before and after rimiducid, including samples of the CNS for PK analysis if |
| | the patient's condition allows. If there is evidence improvement (e.g. partial |
| | response) but not complete resolution after the first dose of rimiducid, then |
| | rimiducid can be repeated every 48 hours for up to 3 doses. Please notify the |
| | medical monitor at Bellicum prior to the administration of rimiducid for<br>neurotoxicity. |
| | <ul> <li>Peripheral blood should be evaluated for BPX-501 cells (CD3+CD19+) at</li> </ul> |
| | the following times: |
| | o Prior to administration of systemic corticosteroid doses (e.g, |
| | methylprednisolone), at 4 and 24 hours (± 30 minutes) post- |
| | systemic corticosteroid doses, and at 7, 14, 21 and 28 days (± 24 |
| | hours) post-systemic corticosteroid doses |
| | <ul> <li>Within 4 hours (± 30 minutes) prior to initiation of rimiducid<br/>infusion, 30 minutes (± 5 minutes) after initiation of infusion, at 2</li> </ul> |
| | hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours (± 30 minutes) |
| | (split samples). Subsequently at 48 hours (± 30 minutes), 7 days |
| | (after initiation of infusion of each dose of rimiducid), and at 14 |
| | days, 21 days, and 28 days (± 24 hours) after the final dose of |
| | rimiducid (if more than one dose is administered) blood samples |
| | will be drawn. Vital signs are recorded prior to rimiducid, and 15, |
| | 30, 60, 120 and 240 minutes (± 5 minutes) after start of infusion. |
| | o If cerebrospinal fluid (CSF) can be safely obtained, CSF should be |
| | sent to the Sponsor for research use to evaluate for BPX-501 cells (CD3+CD19+) prior to initiation of high-dose corticosteroids or |
| | rimiducid. If a sample of CSF can be safely obtained after initiation |


| | of corticosteroids and/or rimiducid for the treatment of |
|---|---|
| | neurotoxicity, CSF should be sent to the Sponsor for research use to |
| | evaluate for BXP-501 cells (CD3+CD19+) (see Table E.3) |
| Grade ≥ 2 | Perform routine institutional care for patients with altered mental |
| (Generalized) <sup>2</sup> | status/obtundation (eg, continuous vital sign monitoring, oxygen, suction, airway protection measurements and consideration of need for mechanical ventilation, ICU admission) |
| | Neurology consult and EEG evaluation |
| | CBC analysis and peripheral blood smear evaluation to evaluate for |
| | thrombotic microangiopathy (TTP/HUS) |
| | <ul> <li>Evaluation for electrolyte and acid-base etiologies</li> </ul> |
| | <ul> <li>Evaluation for liver dysfunction and evidence of hyperammonemia/veno-<br/>occlusive disease (VOD)</li> </ul> |
| | Perform daily neurological and mini-mental status examinations during |
| | hospitalizations to evaluate for resolution/worsening of symptoms |
| | <ul> <li>Perform CNS imaging (MRI and/or contrast enhanced CT)</li> <li>Perform CSF evaluation for presence of cell counts (and differential),</li> </ul> |
| | glucose, protein and gram stain for bacteria. |
| | CSF evaluations for other infectious etiologies (eg, herpes viruses, JC virus, fungal, West Nile virus and toxoplasma) CSF samples should be sent to the Sponsor for research use to |
| | evaluate for the presence of BPX-501 cells |
| | <ul> <li>Consider empiric use of anticonvulsants if seizure is expected</li> </ul> |
| | o Special consideration should be considered for conditioning agents |
| | (eg, Busulfan) or prophylactic GVHD medications (eg, calcineurin inhibitors) as an etiology and institutional guidelines should be instituted for possible treatments (eg, prophylactic GVHD |
| | <ul> <li>medication changes and/or treatment with seizure medications)</li> <li>Consideration of high-dose corticosteroid treatment (1000 mg/day x 3-5 days for adults or 30 mg/kg/day x 2-5 days in children) if no evidence of CNS/systemic infection</li> </ul> |
| | Consideration of empiric antiviral and/or anti-fungal therapy as per institutional standard of care should be considered if infectious etiology is suspected (tailored for lab data results) |
| | A brain biopsy should be considered if other diagnostic tests are unrevealing as to an etiology. |
| | <ul> <li>Rimiducid may be administered if CNS infection ruled out and no<br/>improvement after 48 hours of high-dose corticosteroids (1000 mg/day x 2<br/>days for adults or 30 mg/kg/day x 2 days in children) rimiducid may be<br/>administered in conjunction with corticosteroids and anti-infective agents.<br/>Samples for PK analysis of rimiducid for research use, should be collected<br/>before and after rimiducid, including samples of the CNS for PK analysis if</li> </ul> |
| | the patient's condition allows. If there is evidence improvement (e.g. partial response) but not complete resolution after the first dose of rimiducid, then rimiducid can be given every 48 hours for 3 doses. Please notify the medical monitor at Bellicum prior to the administration of rimiducid for |
| | neurotoxicity. |
| | <ul> <li>Peripheral blood will be collected for research purposes to evaluate BPX-<br/>501 cells (CD3+CD19+) at the following times:</li> </ul> |
| | o Prior to administration of systemic corticosteroid doses (e.g., |
| | methylprednisolone), at 4 and 24 hours (± 30 minutes) post- |
| | systemic corticosteroid doses, and at 7, 14, 21 and 28 days (± 24 |
| | hours) post-systemic corticosteroid doses |
| | <ul> <li>Within 4 hours (± 30 minutes) prior to initiation of rimiducid<br/>infusion, 30 minutes (± 5 minutes) after initiation of infusion, at 2</li> </ul> |


hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours ( $\pm$  30 minutes) (split samples), and subsequently at 48 hours ( $\pm$  30 minutes), and 7 days ( $\pm$  24 hours) (after initiation of infusion of each dose of rimiducid), and at 14 days, 21 days, and 28 days ( $\pm$  30 minutes) after the final dose of rimiducid (if more than one dose is administered) blood samples will be drawn. Vital signs are recorded prior to rimiducid, and 15, 30, 60, 120 and 240 minutes ( $\pm$  5 minutes) after start of infusion.

 If cerebrospinal fluid (CSF) can be safely obtained, CSF should be sent to Sponsor for research use to evaluate for BPX-501 cells (CD3+CD19+) prior to initiation of high-dose corticosteroids or rimiducid. If a sample of CSF can be safely obtained after initiation of corticosteroids and/or rimiducid for the treatment of neurotoxicity, CSF should be sent to the Sponsor for research use to evaluate for BXP-501 cells (CD3+CD19+) (see Table E.3)

http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc htm#ctc 40

- Includes but not limited to cranial nerve abnormalities, brachial plexopathy, ischemia, nystagmus, pyramidal tract syndrome, radiculitis, focal seizure, stroke, transient ischemic attack
- Includes but not limited to aphonia, ataxia, cognitive disturbance, depressed level of consciousness, dysarthria, dysphasia, encephalopathy, headache, hypersomnia, lethargy, memory impairment, meningismus, seizures, somnolence, tremor, visual disturbances

Table E.3: Recommended Procedures to Rule-out Contraindications for LP and Procedures to Minimize Risks\*

| | to Minimize Risks | |
|---|---|---|
| Recomm | ended Procedures | Risk Factors |
| Rule out I | LP contraindication | Coagulopathy |
| 1. B | Brain imaging before LP in case of: | Uncorrected bleeding diathesis |
| | <ul> <li>an intracranial lesion with mass effect</li> </ul> | 100 |
| | <ul> <li>abnormal intracranial pressure</li> </ul> | Anti-coagulant medication |
| | <ul> <li>c. tonsillar herniation is suspected</li> </ul> | |
| | d. recent seizures | |
| | <ul> <li>e. impaired consciousness</li> </ul> | |
| | f. papilledema | |
| | theck platelet and coagulation status (platelet > 40 X | |
| 10 | 0 <sup>9</sup> /L; INR <1.5) | |
| 3. C | theck medications before LP | |
| Patient-rel | lated risk factors: | |
| • D | Determine risk profile and inform patient before and | |
| dı | uring LP procedure | |
| Procedure | es to Minimize Risk | |
| 1. 2: | 5G atraumatic needle; small needle/atraumatic | Post-LP Headache, back pain, post-LP |
| ne | eedle | complaints, |
| | 4 LP attempts | |
| 3. P | assive withdrawal | |
| 4. L | ateral recumbent position | |
| 1. C | Collections up to 30 mL | |

#### References:

de Brabander C, et al. Increased incidence of neurological complications in patients receiving an allogeneic bone marrow transplantation from alternative donors. J Neurol Neurosurg Psychiatry. 2000,68:36-40.

Dowling MR, et al. Neurologic complications after allogeneic hematopoietic stem cell transplantation: risk factors and impact. Bone Marrow Transplantation 2017;1-8.

Folstein MF, et al. "Mini-mental state": a practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res 1975:12:189-198.

Mental Status Examination in Primary Care: A Review. American Family Physician. 2009:80: No.8. pp809-814.
Syed FI CNS complications of hematopoietic stem cell transplant. Hematol Oncol Clin N Am 2016, 30:887-898.
Uckan D, Life-threatening neurological complications after bone marrow transplantation. BMT 2005, 35:71-76.


<sup>\*</sup> All grading corresponding to NCI CTCAE v4.03:





Triplicate ECG: at pre-dose only.

Taken ~5 min prior to blood draws.



ECG: Should be taken ~5 min prior to blood draws.





2 hr sample must be taken  $\leq$  5 min prior to end of rimiducid infusion.



Cellular Kinetics Sample.

| Assessments: GVHD Treatment with rimiducid | | | |
|---|---|---|---|
| Time Point <sup>1</sup> | BPX-501 Cellular Kinetics<br>(CD3+/ CD19+) | Rimiducid PK (plasma) | ECG <sup>4</sup> |
| Pre-Dose (≤ 4 hr) | <b>✓</b> | <b>✓</b> | √ (triplicate) |
| 30 minutes | ✓ | <b>✓</b> | ✓ |
| 2 hr | √2 | √2 | <b>√</b> |
| 4 hr | ✓ | ✓ | ✓ |
| 6 hr | ✓ | ✓ | ✓ |
| 8 hr | ✓ | <b>√</b> | ✓ |
| 12 hr | <b>√</b> | <b>✓</b> | ✓ |
| 24 hr | ✓ | ✓ | ✓ |
| 48 hr | ✓ | N/A | N/A |
| 7 days | ✓ | N/A | N/A |
| 14 days | √3 | N/A | N/A |
| 21 days | √3 | N/A | N/A |
| 28 days | √3 | N/A | N/A |

<sup>&</sup>lt;sup>1</sup>Rimiducid is infused over 2 hours. The reference point for all time points (0 hr) is the initiation of the rimiducid infusion.


<sup>&</sup>lt;sup>2</sup>The 2 hr PK must be collected ≤ 5 min prior to the end of the rimiducid infusion.

After the last dose of rimiducid

<sup>&</sup>lt;sup>4</sup> All ECG should be performed approximately ≤ 5 mins prior to any sample collection if there is a collection at the same time-point.